CLINICAL TRIAL: NCT06249074
Title: The Impact of Gluten-free Diet on the Thyroid Function, Quality of Life and Gut Microbiome Composition in Women With Autoimmune Thyroiditis
Brief Title: Gluten-free Diet in Women With Autoimmune Thyroiditis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Gdansk (Other)
Collaborators: Nutricia Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: RG 4/2020
Record Dates: First submitted 2024-01-31; First posted 2024-02-08 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-01

CONDITIONS: Autoimmune Thyroiditis
Keywords: diet; gut microbiome; thyroid; gluten-free diet
MeSH Terms: conditions — Thyroiditis, Autoimmune; Thyroid Diseases | interventions — Diet, Gluten-Free; Glutens; Dietary Supplements

STUDY DESIGN:
Intervention Model Description: All participants followed normocaloric gluten-free diet for 8 weeks. After first 4 weeks participants were randomly assigned to one of two groups. One group over next 4 weeks additionally to gluten-free diet received gluten in gastrosoluble capsules and second group - rice starch (placebo).
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gluten (Experimental): Gluten group received gluten in gastrosoluble capsules - 2 g of gluten in 3 capsules daily for 4 weeks (week 5 to week 8).
  Interventions: Other: Gluten-free diet; Other: Gluten capsules supplementation
- Placebo (Placebo Comparator): Placebo group received rice starch in gastrosoluble capsules - 3 capsules daily for 4 weeks (week 5 to week 8).
  Interventions: Other: Gluten-free diet; Other: Placebo capsules supplementation

INTERVENTIONS:
Other: Gluten-free diet — Diet with gluten elimination followed by all participants for 8 weeks
Other: Gluten capsules supplementation — 2 g of gluten given in 3 capsules daily for 4 weeks (week 5 to week 8)
  Arms: Gluten
Other: Placebo capsules supplementation — Rice starch in gastrosoluble capsules given in 3 capsules daily for 4 weeks (week 5 to week 8).
  Arms: Placebo

SUMMARY:
The purpose of this interventional study was to check if the elimination of gluten from the diet of women with autoimmune thyroiditis affects their health and thyroid function, quality of life, and the gut microbiome composition.

The main questions it aimed to answer were:

* Does the gluten-free diet worsen the gut microbiome composition?
* Does the gluten-free diet improve thyroid function, measured as thyroid stimulating hormone (TSH), thyroid hormones thyroxine (FT4) and triiodothyronine (FT3), thyroid peroxidase antibodies (TPOAb) and thyroglobulin antibodies (TgAb)?
* Does the gluten-free diet improve the quality of life?

Participants:

* followed normocaloric gluten-free diet for 8 weeks
* after first 4 weeks were randomly assigned to one of two groups. One group over next 4 weeks additionally to gluten-free diet received gluten in gastrosoluble capsules and second group - rice starch (placebo).

Blood and stool samples were collected before diet (T0), after 4 weeks (T1) and after 8 weeks of diet (T2) (total of 3 samples per participant). Also each participant completed the ThyPROpl quality of life assessment questionnaire for patients with thyroid diseases in three time points: before the diet (T0), after 4 weeks (T1) and after 8 weeks of the diet (T2).

ELIGIBILITY:
Inclusion Criteria:

* autoimmune thyroiditis diagnosed by endocrinologist based on increased TPOAb and/or TgAb levels;
* stabilized thyroid function, i.e. thyroid hormones within normal range;
* BMI indicating correct body mass, i.e. within 18.5 - 24.9 kg/m^2.

Exclusion Criteria:

* newly diagnosed autoimmune thyroiditis and unregulated thyroid hormones (hypothyroidism or hyperthyroidism);
* concomitant celiac disease and / or wheat allergy;
* gluten-free diet followed during 6 months prior to enrollment;
* intestinal disorders;
* antibiotic or probiotic therapy during 6 months prior to enrollment.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only women were included in the study because they are much more likely to suffer from autoimmune thyroiditis and to ensure more uniform results in the selected age group.
Enrollment: 31 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2021-11-16 (Actual); Study Completion 2021-11-30 (Actual)

PRIMARY OUTCOMES:
Change in gut microbiome composition | Baseline (T0) to week 4 (T1)
  Bacterial DNA was extracted from stool samples and then 16S rRNA sequencing was conducted to check the change in presence of various bacterial taxa.
Change in gut microbiome composition | Week 4 (T1) to week 8 (T2)
  Bacterial DNA was extracted from stool samples and then 16S rRNA sequencing was conducted to check the change in presence of various bacterial taxa.
Change in thyroid stimulating hormone (TSH) | Baseline (T0) to week 4 (T1)
Change in thyroid stimulating hormone (TSH) | Week 4 (T1) to week 8 (T2)
Change in thyroid hormone thyroxine (FT4) | Baseline (T0) to week 4 (T1)
Change in thyroid hormone thyroxine (FT4) | Week 4 (T1) to week 8 (T2)
Change in thyroid hormone triiodothyronine (FT3) | Baseline (T0) to week 4 (T1)
Change in thyroid hormone triiodothyronine (FT3) | Week 4 (T1) to week 8 (T2)
Change in thyroid peroxidase antibodies (TPOAb) | Baseline (T0) to week 4 (T1)
Change in thyroid peroxidase antibodies (TPOAb) | Week 4 (T1) to week 8 (T2)
Change in thyroglobulin antibodies (TgAb) | Baseline (T0) to week 4 (T1)
Change in thyroglobulin antibodies (TgAb) | Week 4 (T1) to week 8 (T2)
Change in quality of life measured in ThyPROpl questionnaire | Baseline (T0) to week 4 (T1)
  ThyPROpl is a linguistically validated version of the original ThyPRO questionnaire. ThyPRO is recommended for the assessment of health-related quality of life in patients with benign thyroid disease.
  ThyPRO consists of 85 questions summarised in 13 scales measuring aspects of QoL relevant to thyroid patients. Patients are asked to rate their responses for each item on a five-point Likert scale: 0 - not at all; 1 - a little; 2 - some; 3 - quite a bit; 4 - very much. Higher scores mean an improvement in the quality of life.
Change in quality of life measured in ThyPROpl questionnaire | Week 4 (T1) to week 8 (T2)
  ThyPROpl is a linguistically validated version of the original ThyPRO questionnaire. ThyPRO is recommended for the assessment of health-related quality of life in patients with benign thyroid disease.
  ThyPRO consists of 85 questions summarised in 13 scales measuring aspects of QoL relevant to thyroid patients. Patients are asked to rate their responses for each item on a five-point Likert scale: 0 - not at all; 1 - a little; 2 - some; 3 - quite a bit; 4 - very much. Higher scores mean an improvement in the quality of life.

SECONDARY OUTCOMES:
Change in erythrocyte sedimentation rate (ESR) | Baseline (T0) to week 4 (T1)
Change in erythrocyte sedimentation rate (ESR) | Week 4 (T1) to week 8 (T2)
Change in C-reactive protein (CRP) | Baseline (T0) to week 4 (T1)
Change in C-reactive protein (CRP) | Week 4 (T1) to week 8 (T2)
Change in fasting glucose | Baseline (T0) to week 4 (T1)
Change in fasting glucose | Week 4 (T1) to week 8 (T2)

CONTACTS AND LOCATIONS:
Overall Officials: Aleksandra Rodziewicz, MSc, Principal Investigator — Medical University of Gdansk
Locations (1):
- Medical University of Gdańsk, Gdansk, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McGrogan A, Seaman HE, Wright JW, de Vries CS. The incidence of autoimmune thyroid disease: a systematic review of the literature. Clin Endocrinol (Oxf). 2008 Nov;69(5):687-96. doi: 10.1111/j.1365-2265.2008.03338.x. Epub 2008 Jul 31. PMID 18673466
- [Result] Caturegli P, Kimura H, Rocchi R, Rose NR. Autoimmune thyroid diseases. Curr Opin Rheumatol. 2007 Jan;19(1):44-8. doi: 10.1097/BOR.0b013e3280113d1a. PMID 17143095
- [Result] McLeod DS, Cooper DS. The incidence and prevalence of thyroid autoimmunity. Endocrine. 2012 Oct;42(2):252-65. doi: 10.1007/s12020-012-9703-2. Epub 2012 May 29. PMID 22644837
- [Result] Vanderpump MP. The epidemiology of thyroid disease. Br Med Bull. 2011;99:39-51. doi: 10.1093/bmb/ldr030. PMID 21893493
- [Result] Proal AD, Albert PJ, Marshall TG. The human microbiome and autoimmunity. Curr Opin Rheumatol. 2013 Mar;25(2):234-40. doi: 10.1097/BOR.0b013e32835cedbf. PMID 23370376
- [Result] Ishaq HM, Mohammad IS, Guo H, Shahzad M, Hou YJ, Ma C, Naseem Z, Wu X, Shi P, Xu J. Molecular estimation of alteration in intestinal microbial composition in Hashimoto's thyroiditis patients. Biomed Pharmacother. 2017 Nov;95:865-874. doi: 10.1016/j.biopha.2017.08.101. Epub 2017 Sep 10. PMID 28903182
- [Result] Wu GD, Chen J, Hoffmann C, Bittinger K, Chen YY, Keilbaugh SA, Bewtra M, Knights D, Walters WA, Knight R, Sinha R, Gilroy E, Gupta K, Baldassano R, Nessel L, Li H, Bushman FD, Lewis JD. Linking long-term dietary patterns with gut microbial enterotypes. Science. 2011 Oct 7;334(6052):105-8. doi: 10.1126/science.1208344. Epub 2011 Sep 1. PMID 21885731
- [Result] De Filippis F, Pellegrini N, Vannini L, Jeffery IB, La Storia A, Laghi L, Serrazanetti DI, Di Cagno R, Ferrocino I, Lazzi C, Turroni S, Cocolin L, Brigidi P, Neviani E, Gobbetti M, O'Toole PW, Ercolini D. High-level adherence to a Mediterranean diet beneficially impacts the gut microbiota and associated metabolome. Gut. 2016 Nov;65(11):1812-1821. doi: 10.1136/gutjnl-2015-309957. Epub 2015 Sep 28. PMID 26416813
- [Result] Krysiak R, Szkrobka W, Okopien B. The Effect of Gluten-Free Diet on Thyroid Autoimmunity in Drug-Naive Women with Hashimoto's Thyroiditis: A Pilot Study. Exp Clin Endocrinol Diabetes. 2019 Jul;127(7):417-422. doi: 10.1055/a-0653-7108. Epub 2018 Jul 30. PMID 30060266
- [Result] Poblocki J, Panka T, Szczuko M, Telesinski A, Syrenicz A. Whether a Gluten-Free Diet Should Be Recommended in Chronic Autoimmune Thyroiditis or Not?-A 12-Month Follow-Up. J Clin Med. 2021 Jul 22;10(15):3240. doi: 10.3390/jcm10153240. PMID 34362024
- [Result] Ch'ng CL, Jones MK, Kingham JG. Celiac disease and autoimmune thyroid disease. Clin Med Res. 2007 Oct;5(3):184-92. doi: 10.3121/cmr.2007.738. PMID 18056028
- [Result] Roy A, Laszkowska M, Sundstrom J, Lebwohl B, Green PH, Kampe O, Ludvigsson JF. Prevalence of Celiac Disease in Patients with Autoimmune Thyroid Disease: A Meta-Analysis. Thyroid. 2016 Jul;26(7):880-90. doi: 10.1089/thy.2016.0108. PMID 27256300
- [Result] Sanz Y. Effects of a gluten-free diet on gut microbiota and immune function in healthy adult humans. Gut Microbes. 2010 May-Jun;1(3):135-7. doi: 10.4161/gmic.1.3.11868. Epub 2010 Mar 16. PMID 21327021
- [Result] Nistal E, Caminero A, Vivas S, Ruiz de Morales JM, Saenz de Miera LE, Rodriguez-Aparicio LB, Casqueiro J. Differences in faecal bacteria populations and faecal bacteria metabolism in healthy adults and celiac disease patients. Biochimie. 2012 Aug;94(8):1724-9. doi: 10.1016/j.biochi.2012.03.025. Epub 2012 Apr 20. PMID 22542995
- [Result] Di Sabatino A, Volta U, Salvatore C, Biancheri P, Caio G, De Giorgio R, Di Stefano M, Corazza GR. Small Amounts of Gluten in Subjects With Suspected Nonceliac Gluten Sensitivity: A Randomized, Double-Blind, Placebo-Controlled, Cross-Over Trial. Clin Gastroenterol Hepatol. 2015 Sep;13(9):1604-12.e3. doi: 10.1016/j.cgh.2015.01.029. Epub 2015 Feb 19. PMID 25701700
- [Result] Ley RE, Turnbaugh PJ, Klein S, Gordon JI. Microbial ecology: human gut microbes associated with obesity. Nature. 2006 Dec 21;444(7122):1022-3. doi: 10.1038/4441022a. PMID 17183309
- [Result] El-Zawawy HT, Ahmed SM, El-Attar EA, Ahmed AA, Roshdy YS, Header DA. Study of gut microbiome in Egyptian patients with autoimmune thyroid diseases. Int J Clin Pract. 2021 May;75(5):e14038. doi: 10.1111/ijcp.14038. Epub 2021 Feb 4. PMID 33482041
- [Result] Cayres LCF, de Salis LVV, Rodrigues GSP, Lengert AVH, Biondi APC, Sargentini LDB, Brisotti JL, Gomes E, de Oliveira GLV. Detection of Alterations in the Gut Microbiota and Intestinal Permeability in Patients With Hashimoto Thyroiditis. Front Immunol. 2021 Mar 5;12:579140. doi: 10.3389/fimmu.2021.579140. eCollection 2021. PMID 33746942
- [Result] Zhao F, Feng J, Li J, Zhao L, Liu Y, Chen H, Jin Y, Zhu B, Wei Y. Alterations of the Gut Microbiota in Hashimoto's Thyroiditis Patients. Thyroid. 2018 Feb;28(2):175-186. doi: 10.1089/thy.2017.0395. Epub 2018 Feb 1. PMID 29320965
- [Result] Xu Q, Ni JJ, Han BX, Yan SS, Wei XT, Feng GJ, Zhang H, Zhang L, Li B, Pei YF. Causal Relationship Between Gut Microbiota and Autoimmune Diseases: A Two-Sample Mendelian Randomization Study. Front Immunol. 2022 Jan 24;12:746998. doi: 10.3389/fimmu.2021.746998. eCollection 2021. PMID 35140703
- [Result] Bonder MJ, Tigchelaar EF, Cai X, Trynka G, Cenit MC, Hrdlickova B, Zhong H, Vatanen T, Gevers D, Wijmenga C, Wang Y, Zhernakova A. The influence of a short-term gluten-free diet on the human gut microbiome. Genome Med. 2016 Apr 21;8(1):45. doi: 10.1186/s13073-016-0295-y. PMID 27102333
- [Result] De Palma G, Nadal I, Collado MC, Sanz Y. Effects of a gluten-free diet on gut microbiota and immune function in healthy adult human subjects. Br J Nutr. 2009 Oct;102(8):1154-60. doi: 10.1017/S0007114509371767. Epub 2009 May 18. PMID 19445821